CLINICAL TRIAL: NCT04209985
Title: Reaching for Equity in Sleep Apnea Treatment (REST): Pilot of Telephonic Health Coaching Intervention to Improve Adherence to Sleep Apnea Treatment
Brief Title: Reaching for Equity in Sleep Apnea Treatment (REST) Study
Acronym: REST pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-27249
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Sleep Apnea
Keywords: Health coaching; Adherence to treatment; Health disparities
MeSH Terms: conditions — Sleep Apnea Syndromes; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: Patients are randomly assigned to receive health coaching or usual care. Patients assigned to usual care have access to all existing resources, including technical support from durable medical equipment providers, respiratory therapist visits with the Sleep Clinic, group visits, or visits with their primary care provider. Patients in the health coaching arm have access to all usual care resources. In addition, they will be assigned an unlicensed, trained health coach who will call them up to five times to identify and resolve barriers to adherence, including lack of understanding of their condition or the treatment, discomfort in acclimating to treatment, technical difficulties in mask fit or device settings, and challenges in navigating durable medical equipment providers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health coaching arm (Experimental): For the health coaching arm, an unlicensed, trained health coach will call patients up to five times to identify and resolve barriers to adherence, including lack of understanding of their condition or the treatment, discomfort in acclimating to treatment, technical difficulties in mask fit or device settings, and challenges in navigating durable medical equipment providers.
  Interventions: Behavioral: Health coaching
- Usual care (No Intervention): Patients assigned to usual care have access to all other available resources, including technical support from durable medical equipment providers, respiratory therapist visits with the Sleep Clinic, group visits, or visits with their primary care provider.

INTERVENTIONS:
Behavioral: Health coaching — Brief telephonic intervention consisting of up to five phone calls from a health coach
  Arms: Health coaching arm

SUMMARY:
This study will test a brief telephonic health coaching intervention to improve adherence to positive airway pressure therapy for treatment of obstructive sleep apnea.

DETAILED DESCRIPTION:
The investigators will carry out a pilot study in which patients will be randomly assigned to receive health coaching or usual care. Participants are English- and Spanish-speaking patients from a county-based public health system who have received a positive airway pressure device for the treatment of sleep apnea. An unlicensed, trained health coach will call patients three times to resolve barriers to adherence. Primary outcomes include both adherence measures collected by the device modem at baseline and 4 months, and patient-reported outcomes such as daytime sleepiness.

ELIGIBILITY:
Inclusion Criteria:

* English- or Spanish-speaking
* At least 18 years of age
* Had previously received a modem-enabled positive airway pressure device for the treatment of sleep apnea
* Not currently meeting Medicare standards for adherence of at least 4 hours per night for at least 70% of the last 30 nights
* Received care from the San Francisco General Hospital Sleep Clinic

Exclusion Criteria:

* Not English- or Spanish-speaking
* Younger than 18 years
* Does not have phone number at which could be reached

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-11-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean number of hours used on average over the last 30 days | Enrollment to 4 months post enrollment
  Total number of hours PAP device used during 30 day period divided by 30 days (PAP device is part of existing clinical care)

SECONDARY OUTCOMES:
Proportion using device at any time in last 30 days | Enrollment to 4 months post enrollment
  Numerator: Number of people using PAP device at any time in last 30 days; Denominator: Number of people in study arm (PAP device is part of existing clinical care)
Patient-reported daytime sleepiness | Enrollment to 4 months post enrollment
  Mean score on the Epworth Sleepiness Scale (8 items with aggregate scale of 0-24 points, where 24 indicates greatest sleepiness symptoms)
Attitudes to PAP treatment | Enrollment to 4 months post enrollment
  Mean score on the Attitudes to PAP Treatment Inventory (5 items with combined scale of 4-25, where higher scores indicate negative attitudes toward PAP treatment)
Confidence in using PAP therapy | Enrollment to 4 months post enrollment
  Mean score on self-efficacy for use of PAP therapy (4 items, with combined scale from 0-40, where 40 indicates greatest self-efficacy)
Mean number of hours used on average over the last 30 days on nights that device was used | Enrollment to 4 months post enrollment
  Total number of hours device used during 30 day period divided by the number of days on which the device was used
Mean proportion of last 30 days in which device used at least 4 hours/night | Enrollment to 4 months post enrollment
  Mean across group of: (Numerator: Number of days in last 30 days that PAP device was used at least 4 hours; Denominator: 30 days) (PAP device is part of existing clinical care)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Willard-Grace, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital Sleep Clinic, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No